CLINICAL TRIAL: NCT02576054
Title: A Phase III, Open-Label, Clinical Trial to Study the Safety and Immunogenicity of the Quadrivalent HPV (Types 6, 11, 16, 18) L1 VLP Particle (VLP) Vaccine in 9- to 15-Year-Old Japanese Boys
Brief Title: Safety and Tolerability Study of V501 in Japanese Boys (V501-200)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V501-200
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Anogenital Human Papilloma Virus Infection; Condyloma Acuminata
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- V501 (Experimental): 0.5 mL intramuscular injection on Day 1, Month 2, and Month 6
  Interventions: Biological: V501

INTERVENTIONS:
Biological: V501 — Quadrivalent HPV [Type 6, 11, 16 and 18] L1 VLP vaccine), 0.5 mL intramuscular injection on Day 1, Month 2, and Month 6
  Other Names: Gardasil™

SUMMARY:
This is a study of V501 [quadrivalent Human Papillomavirus (HPV) (Type 6, 11, 16 and 18) L1 virus-like particle (VLP) vaccine] in healthy Japanese boys. This study will consist of two periods. Period I of the study is to evaluate the immunogenicity and tolerability of V501 up to Month 7. Period II of the study is to evaluate the long-term immunogenicity and safety from Month 7 to Month 30. Two analyses are planned. The first analysis will be conducted when all subjects have completed their Month 7 visit or have been discontinued before that time. The second analysis will be conducted at the end of study. The primary hypothesis tested in this study is that seroconversion rates for the vaccine HPV types will be >90% at 4 weeks postdose 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male
* Have a legal representative who provides written informed consent for the trial on the participant's behalf
* Have a legal representative who is able to read, understand, and complete the vaccine report card
* Has not yet had coitarche and does not plan on becoming sexually active from Day 1 through Month 7 of the study
* Other inclusion criteria will be discussed with the investigator during screening

Exclusion Criteria:

* Currently enrolled in clinical studies of investigational agents
* History of known prior vaccination with an HPV vaccine or plans to receive one outside the study
* History of severe allergic reaction that required medical intervention
* Allergic to any vaccine component, including aluminum, yeast, or BENZONASE™
* Received immune globulin or blood-derived products in the past 6 months or plans to receive any before Month 7 of the study
* History of splenectomy, is currently immunocompromised, or has been diagnosed with immunodeficiency, Human Immunodeficiency Virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition
* Received immunosuppressive therapy in the past year, excluding inhaled, nasal, or topical corticosteroids
* Known thrombocytopenia or coagulation disorder that would contraindicate intramuscular injections
* Ongoing alcohol or drug abuse within the past 12 months
* History of genital warts or a positive test for HPV

Ages: 9 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- MSD K.K., Chiyoda-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Murata S, Takeuchi Y, Yamanaka K, Hayakawa J, Yoshida M, Yokokawa R, Wakana A, Sawata M, Tanaka Y. Safety and Immunogenicity of the Quadrivalent HPV Vaccine in Japanese Boys: a Phase 3, Open-Label Study. Jpn J Infect Dis. 2019 Sep 19;72(5):299-305. doi: 10.7883/yoken.JJID.2018.448. Epub 2019 May 31. PMID 31155600

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | V501
Started | 101
Vaccination 1 | 100
Vaccination 2 | 100
Vaccination 3 | 100
Completed | 100
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | V501
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 101
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion for HPV Types 6, 11, 16, and 18
Description: Antibodies to HPV Types 6, 11, 16, and 18 were measured using a competitive luminex immunoassay 4 weeks after 3rd vaccination (Month 7). Antibody titers were expressed as milli Merck units/mL (mMU/mL). Seroconversion was defined as an anti-HPV 6 titer ≥20 mMU/mL, an anti-HPV 11 titer ≥16 mMU/mL, an anti-HPV 16 titer of ≥20 mMU/mL and an anti-HPV 18 titer of ≥24 mMU/mL.
Time Frame: Four weeks postdose 3 (Month 7)
Population: All participants that received all 3 vaccinations within acceptable day ranges, were seronegative to the relevant HPV type at Day 1, did not have protocol violations that could interfere with evaluation of the immune response, and provided Month 7 serology result within 21 to 49 days post dose 3.
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V501
Number analyzed (Participants) | 99
Percentage of Participants
  Anti HPV 6: number analyzed (Participants) | 98
  Anti HPV 6 | 94.9 [88.5 to 98.3]
  Anti HPV 11: number analyzed (Participants) | 98
  Anti HPV 11 | 99.0 [94.4 to 100.0]
  Anti HPV 16 | 99.0 [94.5 to 100.0]
  Anti HPV 18: number analyzed (Participants) | 98
  Anti HPV 18 | 99.0 [94.4 to 100.0]

2. Primary Outcome: Percentage of Participants With Elevated Oral Temperature (>=37.5° C)
Description: The parent/guardian of the participant was to record the participant's oral temperature in the evening after each study vaccination and daily for 4 days after each study vaccination. Elevated temperature was defined as ≥99.5°F (≥37.5ºC). The percentage of participants that had an elevated temperature was summarized.
Time Frame: Up to Day 5 after any vaccination
Population: All participants who received at least 1 study vaccination and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | V501
Number analyzed (Participants) | 100
Percentage of Participants
  ≥ 37.5 °C (99.5 °F) and < 38.0 °C (100.4 °F) | 3.0
  ≥ 38.0 °C (100.4 °F) and < 38.5 °C (101.3 °F) | 1.0
  ≥ 38.5 °C (101.3 °F) | 2.0

3. Primary Outcome: Percentage of Participants With an Injection-site Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study drug. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug or a protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study drug or protocol-specified procedure is also an AE. The parent/guardian of the participant was to record the presence of any vaccination report card (VRC)-prompted injection-site AEs that occurred in the 5 days after any vaccination. The percentage of participants with an injection-site AE prompted on the VRC (erythema, pain, and swelling) was summarized.
Time Frame: Up to Day 5 after any vaccination
Population: All participants who received at least 1 study vaccination and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | V501
Number analyzed (Participants) | 100
Percentage of Participants | 64.0

4. Primary Outcome: Percentage of Participants With a Systemic Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study drug. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug or a protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study drug or protocol-specified procedure is also an AE. The parent/guardian of the participant was to record the presence of any VRC-prompted systemic AEs that occurred in the 5 days after any vaccination. The percentage of participants with a systemic AE was summarized.
Time Frame: Up to Day 15 after any vaccination
Population: All participants who received at least 1 study vaccination and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | V501
Number analyzed (Participants) | 100
Percentage of Participants | 21.0

5. Primary Outcome: Percentage of Participants With a Serious Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, is a cancer, is an overdose, or is another important medical event. The percentage of participants that experienced 1 or more SAEs was summarized.
Time Frame: Up to Day 15 after any vaccination
Population: All participants who received at least 1 study vaccination and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | V501
Number analyzed (Participants) | 100
Percentage of Participants | 0.0

6. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, is a cancer, is an overdose, or is another important medical event. The percentage of participants that experienced 1 or more SAEs that were considered at least possibly related to the study vaccine was summarized.
Time Frame: Up to 30 months
Population: All participants who received at least 1 study vaccination and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | V501
Number analyzed (Participants) | 100
Percentage of Participants | 0.0

7. Secondary Outcome: Geometric Mean Titers for Serum Anti-HPV Types 6, 11, 16, and 18 Participants Aged 9 to 15 Years Versus Participants Aged 16 to 26 Years
Description: Antibodies to HPV Types 6, 11, 16, and 18 were measured using a competitive luminex immunoassay. Antibody titers were expressed mMU/mL. GMTs obtained for each anti-HPV from this study were compared to each of the ant-HPV GMTs obtained in study V501-122 (NCT NCT01862874) in which Japanese males 16 to 26 years received V501 in the same 3 dose regimen, to test a hypothesis that would demonstrate non-inferiority.
Time Frame: Four weeks postdose 3 (Month 7)
Population: Participants 9 to 15 years old (PN200) or 16 to 26 years old (PN122) that received all 3 vaccinations within acceptable day ranges, were seronegative to the relevant HPV type at Day 1, did not have protocol violations that could interfere with evaluation of the immune response, and provided Month 7 serology result within 21 to 49 days post dose 3.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- Participants Aged 9 to 15 Years (PN200); Participants Aged 16 to 26 Years (PN122): 0.5 mL intramuscular injection on Day 1, Month 2, and Month 6
Arm/Group | Participants Aged 9 to 15 Years (PN200) | Participants Aged 16 to 26 Years (PN122)
Number analyzed (Participants) | 99 | 487
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 98 | 472
  Anti-HPV 6 | 482.9 [351.1 to 664.1] | 385.0 [355.7 to 416.7]
  Anti-HPV 11: number analyzed (Participants) | 98 | 472
  Anti-HPV 11 | 1052.8 [851.3 to 1302.0] | 458.4 [424.8 to 494.7]
  Anti-HPV 16: number analyzed (Participants) | 99 | 465
  Anti-HPV 16 | 3878.3 [2908.5 to 5171.6] | 2294.8 [2110.0 to 2495.7]
  Anti-HPV 18: number analyzed (Participants) | 98 | 487
  Anti-HPV 18 | 1114.5 [871.6 to 1425.1] | 365.4 [327.1 to 408.1]
Statistical Analysis 1: Comparison: Participants Aged 9 to 15 Years (PN200) vs Participants Aged 16 to 26 Years (PN122); Anti-HPV 6; Test type: Non-Inferiority — The statistical criterion for success requires that the lower bound of two-sided 95% confidence interval (CI) of GMT ratio between boys enrolled in V501-200 and men enrolled in the Phase III study V501-122 be greater than 0.5% for each HPV type; p < 0.001, ANOVA; Log-transformed data using an analysis of variance model with a term for age-group; GMT Ratio = 1.25, 95% CI 2-sided [1.00 to 1.57] — GMT Ratio= GMT PN200 divided by GMT PN122
Statistical Analysis 2: Comparison: Participants Aged 9 to 15 Years (PN200) vs Participants Aged 16 to 26 Years (PN122); Anti-HPV 11; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.001, ANOVA; Log-transformed data using an analysis of variance model with a term for age-group; GMT Ratio = 2.30, 95% CI 2-sided [1.89 to 2.78] — GMT Ratio = GMT PN200 divided by GMT PN122
Statistical Analysis 3: Comparison: Participants Aged 9 to 15 Years (PN200) vs Participants Aged 16 to 26 Years (PN122); Anti-HPV 16; Test type: Non-Inferiority — The statistical criterion for success requires that the lower bound of two-sided 95% CI of GMT ratio between boys enrolled in V501-200 and men enrolled in the Phase III study V501-122 be greater than 0.5% for each HPV type; p < 0.001, ANOVA; Log-transformed data using an analysis of variance model with a term for age-group; GMT Ratio = 1.69, 95% CI 2-sided [1.35 to 2.11] — GMT Ratio= GMT PN200 divided by GMT PN122
Statistical Analysis 4: Comparison: Participants Aged 9 to 15 Years (PN200) vs Participants Aged 16 to 26 Years (PN122); Anti-HPV 18; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 3]; p < 0.001, ANOVA; Log-transformed data using an analysis of variance model with a term for age-group; GMT Ratio = 3.05, 95% CI 2-sided [2.33 to 3.99] — GMT Ratio= GMT PN200 divided by GMT PN122

8. Secondary Outcome: Geometric Mean Titers for Serum Anti-HPV Types 6, 11, 16, and 18: Persistence at 18 Months
Description: Antibodies to HPV Types 6, 11, 16, and 18 were measured using a competitive luminex immunoassay. Antibody titers were expressed as mMU/mL.
Time Frame: 12 months postdose 3 (18 months)
Population: All participants that received all 3 vaccinations within acceptable day ranges, were seronegative to the relevant HPV type at Day 1, did not have protocol violations that could interfere with evaluation of the immune response, and provided Month 18 data within an acceptable date range of 12 months postdose 3.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | V501
Number analyzed (Participants) | 99
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 97
  Anti-HPV 6 | 222.0 [181.8 to 271.3]
  Anti-HPV 11: number analyzed (Participants) | 97
  Anti-HPV 11 | 259.9 [210.7 to 320.7]
  Anti-HPV 16: number analyzed (Participants) | 98
  Anti-HPV 16 | 1154.1 [937.3 to 1421.0]
  Anti-HPV 18: number analyzed (Participants) | 97
  Anti-HPV 18 | 212.1 [165.6 to 271.7]

9. Secondary Outcome: Geometric Mean Titers for Serum Anti-HPV Types 6, 11, 16, and 18: Persistence at 30 Months
Description: as for outcome 8
Time Frame: 24 months postdose 3 (30 months)
Population: All participants that received all 3 vaccinations within acceptable day ranges, were seronegative to the relevant HPV type at Day 1, did not have protocol violations that could interfere with evaluation of the immune response, and provided Month 30 data within an acceptable date range of 24 months postdose 3.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | V501
Number analyzed (Participants) | 99
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 98
  Anti-HPV 6 | 177.5 [145.0 to 217.2]
  Anti-HPV 11: number analyzed (Participants) | 98
  Anti-HPV 11 | 181.5 [146.3 to 225.2]
  Anti-HPV 16 | 831.3 [680.7 to 1015.1]
  Anti-HPV 18: number analyzed (Participants) | 98
  Anti-HPV 18 | 144.2 [112.2 to 185.2]

10. Secondary Outcome: Percentage of Participants With Seroconversion for HPV Types 6, 11, 16, and 18: Persistence at 18 Months
Description: Serum antibodies to HPV types were measured with a competitive luminex immunoassay. The serostatus cutoffs (mMU/mL) for HPV types were as follows: HPV Type 6: ≥20; HPV Type 11: ≥16; HPV Type 16: ≥20; HPV Type 18: ≥24
Time Frame: 12 months postdose 3 (18 months)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V501
Number analyzed (Participants) | 99
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 97
  Anti-HPV 6 | 97.9 [92.7 to 99.7]
  Anti-HPV 11: number analyzed (Participants) | 97
  Anti-HPV 11 | 100.0 [96.3 to 100.0]
  Anti-HPV 16: number analyzed (Participants) | 98
  Anti-HPV 16 | 99.0 [94.4 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 97
  Anti-HPV 18 | 94.8 [88.4 to 98.3]

11. Secondary Outcome: Percentage of Participants With Seroconversion for HPV Types 6, 11, 16, and 18: Persistence at 30 Months
Description: as for outcome 10
Time Frame: 24 months postdose 3 (30 months)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V501
Number analyzed (Participants) | 99
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 98
  Anti-HPV 6 | 98.0 [92.8 to 99.8]
  Anti-HPV 11: number analyzed (Participants) | 98
  Anti-HPV 11 | 98.0 [92.8 to 99.8]
  Anti-HPV 16 | 99.0 [94.5 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 98
  Anti-HPV 18 | 93.9 [87.1 to 97.7]

ADVERSE EVENTS:
Time Frame: Up to 30 months
Description: Population included all participants that received at least 1 vaccination
Arm/Group | V501
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 67/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V501 (N=100)
Injection site erythema (General disorders) | 31 (57)
Injection site pain (General disorders) | 57 (130)
Injection site pruritus (General disorders) | 6 (10)
Injection site swelling (General disorders) | 34 (63)
Pyrexia (General disorders) | 6 (8)
Nasopharyngitis (Infections and infestations) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT02576054/Prot_SAP_000.pdf